CLINICAL TRIAL: NCT00252642
Title: The Impact of Peginterferon Alpha-2a Maintenance Therapy on Portal Hypertension in Patients With Chronic Hepatitis C Virus Infection and Advanced Fibrosis and Cirrhosis Enrolled in the HALT-C Trial
Brief Title: Peginterferon Alpha-2a Maintenance Therapy for Portal Hypertension in Patients With Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PH-VCU-05
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C; Cirrhosis; Fibrosis
Keywords: Hepatitis C; Interferon; Cirrhosis; Liver Disease; Portal Hypertension; Portal Pressure
MeSH Terms: conditions — Hepatitis C; Fibrosis; Liver Diseases; Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Peginterferon Alpha-2a

SUMMARY:
The primary purpose of this study is to determine if peginterferon alpha-2a maintenance therapy (90 mcg/week) will lower portal pressure in patients with hepatitis C virus infections and advanced fibrosis or cirrhosis.

DETAILED DESCRIPTION:
Portal hypertension develops in patients with advanced fibrosis and cirrhosis and is the primary driving force leading to complications of cirrhosis, hepatic decompensation and mortality in patients with chronic liver disease. None of the three major complications of advanced liver disease variceal hemorrhage, ascites and hepatic encephalopathy occur in the absence of portal hypertension. As a result, measuring portal pressure and treating portal hypertension is an important part in the management of patients with advanced liver disease. A sub-study to measure portal pressure was initially proposed as part of the HALT-C clinical trial. Unfortunately, only 2/10 centers elected to participate in this sub-study and as a result, this was eventually dropped as a sub-study within the HALT-C trial.

Recent data has suggested that interferon therapy may selectively reduce portal hypertension in patients with cirrhosis. In an abstract presented at the 2004 annual meeting of the European Association for the Study of the Liver (EASL), portal pressure declined significantly in patients with NR after 6 months of treatment with peginterferon and ribavirin. At the time portal pressure was measured in this study, a transjugular liver biopsy was also performed to assess the effects of treatment on hepatic histology. Despite a reduction in portal pressure, no reduction in hepatic fibrosis score was observed. This suggested that interferon may reduce portal pressure through a direct affect on the hepatic vasculature; and suggests that interferon may prevent complications of cirrhosis regardless of its effects on HCV RNA and hepatic inflammation. Since portal pressure is the primary factor responsible for complications of cirrhosis including variceal hemorrhage, ascites and hepatic encephalopathy, these preliminary results suggest that maintenance interferon therapy could possibly prevent these complications.

Preliminary results form a randomized, controlled trial of maintenance interferon therapy (Co-Pilot) presented at the 2004 annual meeting of the American Association of the study of Liver Disease (AASLD) did in fact demonstrate that patients with advanced fibrosis or cirrhosis who received maintenance peginterferon maintenance therapy over a two year period had a significant reduction in the incidence of variceal hemorrhage compared to that observed in the control group. The HALT-C trial provides an ideal patient population in which to further assess the effects of maintenance interferon therapy on portal hypertension.

The first patients who were enrolled into the HALT-C trial are scheduled to complete four years of maintenance therapy near the end of 2004. This provides an optimal time point at which to assess the impact of maintenance interferon therapy on portal pressure. Although an ideal study design would have been to measure portal pressure at baseline and then again after 4 years in both the control and treatment groups, measuring portal pressure at the completion of the study will still provide significant information regarding the impact of maintenance interferon therapy on portal hypertension. The number of patients enrolled into HALT-C at these two sites is substantial (nearly 400 patients) and since the control and maintenance therapy groups were well matched at the start of the study we can assume that baseline portal pressure at the time of randomization was not significantly different in the two groups. Thus, if 4 years of maintenance interferon therapy does indeed reduce portal pressure a significant difference in mean portal pressure should be observed between the two groups at the completion of the HALT-C trial.

Patients who were randomized to the control arm of HALT-C during the past four years have received no treatment for chronic HCV during the past 4 years. Such patients will be offered the opportunity to receive peginterferon maintenance therapy for 6 months as part of this protocol and then undergo repeat measurement of portal pressure to determine if they could potentially benefit from remaining on peginterferon maintenance therapy long term

ELIGIBILITY:
Inclusion Criteria:

* Completion of HALT-C Trial, in either treatment or non-treatment arm

Exclusion Criteria:

* Non-completion of HALT-C Trial
* Patients who do not wish to be treated with peginterferon after the first portal pressure measurement
* Hepatocellular Carcinoma
* Underlying autoimmune disorder
* Currently being treated with immune suppressive agent
* Illicit drug use
* Alcohol use of more than 6 grams per day
* Advanced cardiopulmonary disease
* Uncontrolled diabetes mellitus
* Patients who, in the opinion of the investigator, should not participate in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Changes in portal pressure after 6 moths of treatment with peginterferon alfa-2a will be calculated by comparing portal pressure at the end of HALT-C to values obtained after 6 months of peginterferon.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell L. Shiffman, MD, Principal Investigator — Virignia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Alter MJ, Kruszon-Moran D, Nainan OV, McQuillan GM, Gao F, Moyer LA, Kaslow RA, Margolis HS. The prevalence of hepatitis C virus infection in the United States, 1988 through 1994. N Engl J Med. 1999 Aug 19;341(8):556-62. doi: 10.1056/NEJM199908193410802. PMID 10451460
- [Background] Charlton M. Hepatitis C infection in liver transplantation. Am J Transplant. 2001 Sep;1(3):197-203. doi: 10.1034/j.1600-6143.2001.001003197.x. PMID 12102252
- [Background] Poynard T, McHutchison J, Manns M, Trepo C, Lindsay K, Goodman Z, Ling MH, Albrecht J. Impact of pegylated interferon alfa-2b and ribavirin on liver fibrosis in patients with chronic hepatitis C. Gastroenterology. 2002 May;122(5):1303-13. doi: 10.1053/gast.2002.33023. PMID 11984517
- [Background] Imai Y, Kawata S, Tamura S, Yabuuchi I, Noda S, Inada M, Maeda Y, Shirai Y, Fukuzaki T, Kaji I, Ishikawa H, Matsuda Y, Nishikawa M, Seki K, Matsuzawa Y. Relation of interferon therapy and hepatocellular carcinoma in patients with chronic hepatitis C. Osaka Hepatocellular Carcinoma Prevention Study Group. Ann Intern Med. 1998 Jul 15;129(2):94-9. doi: 10.7326/0003-4819-129-2-199807150-00005. PMID 9669992
- [Background] Shiffman ML, Hofmann CM, Contos MJ, Luketic VA, Sanyal AJ, Sterling RK, Ferreira-Gonzalez A, Mills AS, Garret C. A randomized, controlled trial of maintenance interferon therapy for patients with chronic hepatitis C virus and persistent viremia. Gastroenterology. 1999 Nov;117(5):1164-72. doi: 10.1016/s0016-5085(99)70402-6. PMID 10535880
- [Background] Lee WM, Dienstag JL, Lindsay KL, Lok AS, Bonkovsky HL, Shiffman ML, Everson GT, Di Bisceglie AM, Morgan TR, Ghany MG, Morishima C, Wright EC, Everhart JE; HALT-C Trial Group. Evolution of the HALT-C Trial: pegylated interferon as maintenance therapy for chronic hepatitis C in previous interferon nonresponders. Control Clin Trials. 2004 Oct;25(5):472-92. doi: 10.1016/j.cct.2004.08.003. PMID 15465617
- [Background] Garcia N Jr, Sanyal AJ. Portal hypertension. Clin Liver Dis. 2001 May;5(2):509-40. doi: 10.1016/s1089-3261(05)70176-8. PMID 11385974